CLINICAL TRIAL: NCT01634282
Title: A Long-term Clinical Study of OPC-262 in Patients With Type 2 Diabetes on Study (Extension From Study 262-09-001)
Brief Title: Along-term Study of OPC-262 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262-09-002
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-262 (Experimental)
  Interventions: Drug: OPC-262

INTERVENTIONS:
Drug: OPC-262 — Orally administered once daily

SUMMARY:
The purpose of this clinical study is to evaluate the safety of OPC-262 (2.5 mg and 5 mg) in patients with type 2 diabetes by long-term administration orally for 52 weeks and to evaluate the efficacy of OPC-262

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed Study 262-09-001 (namely, patients who visited the hospital at visit Week 24）
* Patients who are capable of giving informed consent prior to participating in this clinical study
* Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner for the entire study period and for 4 weeks after the study (end of the post-observation period)

Exclusion Criteria:

* Patients who withdrew from Study 262-09-001
* Patients who experienced serious adverse events that the relationship with the study drug was not denied in Study 262-09-001
* Patients who experienced serious adverse events that the relationship with the study drug are denied in Study 262-09-001 and whose symptoms are still emerged at the time of initiation of this study
* Patients who met the exclusion criteria of Study 262-09-001 during the study period of Study 262-09-001
* Female patients who wish to become pregnant during the study period of Study 262-09-002 or within 4 weeks after the study
* Patients otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in HBA1c form baseline | 52 Weeks
Incidence and severity of adverse events | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region